CLINICAL TRIAL: NCT06459947
Title: Effect of Cyanoacrylate and Concentrated Growth Factor on Wound Healing and Patient Comfort at the Palatal Donor Site
Brief Title: Effect of Cyanoacrylate and Concentrated Growth Factor on Palatal Donor Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Dicle Altındal, DDS, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 28.02.2024/07
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Wound Healing; Pain; Patient Comfort
Keywords: cyanoacrylate; free gingival graft; concentrated growth factor
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Control group) (Active Comparator): After FGG is taken from the palatal area, the sponge is placed in the wound area.
  Interventions: Procedure: Free gingival graft procedure
- Group 2 (Cyanoacrylate group) (Active Comparator): After the FGG is taken from the palatal area, a cyanoacrylate tissue adhesive is placed in the wound area.
  Interventions: Procedure: Free gingival graft procedure
- Group 3 (Concentrated Growth Factor group) (Active Comparator): After the FGG is taken from the palatal area, concentrated growth factor (CGF) group is placed in the wound area. CGF is obtained by centrifuging blood in four different cycles and times.
  Interventions: Procedure: Free gingival graft procedure

INTERVENTIONS:
Procedure: Free gingival graft procedure — The palatal area is anesthetized using local anesthesia. The free gingival graft (FGG) is taken from the donor site with a scalpel.

SUMMARY:
The aim of this planned randomized controlled clinical study is to evaluate the morbidity of the palatal donor area after free gingival graft (FGG) operations. In this study, wound healing and pain levels in the palatal region will be evaluated after cyanoacrylate and concentrated growth factor (CGF) applications.

DETAILED DESCRIPTION:
Free gingival graft obtained in the palatal region causes morbidity. Therefore, clinicians try to overcome these difficulties by isolating the wound in the palatal region from the oral environment and/or accelerating wound healing.

Periodontal dressings, acrylic stents, hemostatic agents, surgical sponges, platelet concentrates, low-level laser therapy, photobiomodulation, cyanoacrylate tissue adhesives and hyaluronic acid are some of the methods used for donor site management or to accelerate healing.

Cyanoacrylate adhesives form an adhesive film through rapid polymerization triggered by the hydroxyl groups on the surfaces to which they are applied. They have both bacteriostatic and hemostatic properties.

In recent years, it has been observed that the use of platelet concentrates such as Platelet Rich Plasma (PRP), Platelet Rich Fibrin (PRF) and autogenous products such as CGF (concentrated growth factor) in periodontal treatments has increased.

CGF is obtained by centrifuging blood in four different cycles and times. This product contains a relatively intact fibrin clot containing platelets, leukocytes, various growth factors and cytokines. CGF can be applied as a carrier of growth factors and/or a barrier membrane to aid tissue regeneration and wound healing in clinical applications.

The aim of this planned randomized controlled clinical study is to evaluate the morbidity of the palatal donor area after FGG operations. In this study, wound healing and pain levels in the palatal region will be evaluated after cyanoacrylate and CGF applications.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* not had periodontal surgery in the last 6 months

Exclusion Criteria:

* smoker
* allergic to medication
* high anxiety (using modified dental anxiety scale)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-03-02 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
VAS | The pain level is recorded every hour for the first 8 hours after the operation, and on the 2nd, 3rd, 4th, 5th, 6th, 7th days after the operation.
  The patient is given a form to record the post-operative pain level in the palatial area with Visual analogue scale (VAS). The VAS is a scale that rates pain severity from 0 to 10. (0 = no pain to 10 = severe pain)
Epithelialization | The epithelialization is examined on the 7th, 14th, 21st, and 28th days
  Hydrogen peroxide is used to detect epithelialization in the donor area after the operation. If epithelialization is not completed, H2O2 affects the catalase enzyme in the connective tissue and releases water and oxygen. Thus, clinically, it forms blisters on the palatal wound surface. Epithelialization scores will be divided into three groups: absent, partially epitheliazed and completely epithelialized.

SECONDARY OUTCOMES:
Number of analgesic drugs | Number of analgesic drugs is recorded on the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th days.
  Patients are asked to note the number of analgesics they took for pain during the first week.
Healing Index | The Healing Index is recorded on the 7th day.
  The Healing Index is recorded with a 5-level score ranging from 1 (very poor) to 5 (excellent).
Color Match | The color match is evaluated on the 7th, 14th, 21st and 28th days.
  The color match is evaluated by Visual analogue scale (VAS). (0: no color match, 10: perfect color match)
Secondary Bleeding | Post-operative bleeding is recorded on the 1st, 2nd, 3rd, 4th, 5th, 6th, 7th days.
  Post-operative bleeding in the palatal region is noted. The patient notes the postoperative bleeding status of the palatal area. Bleeding scores are recorded as yes or no.

CONTACTS AND LOCATIONS:
Overall Officials: Dicle Altindal, DDS, Principal Investigator — Yuzuncu Yil University; Elif Tore Sari, PhD, Study Chair — Yuzuncu Yil University; Nazli Zeynep Alpaslan, PhD, Study Chair — Yuzuncu Yil University
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lektemur Alpan A, Torumtay Cin G. PRF improves wound healing and postoperative discomfort after harvesting subepithelial connective tissue graft from palate: a randomized controlled trial. Clin Oral Investig. 2020 Jan;24(1):425-436. doi: 10.1007/s00784-019-02934-9. Epub 2019 May 18. PMID 31104113
- [Background] Verissimo AH, Ribeiro AKC, Martins ARLA, Gurgel BCV, Lins RDAU. Comparative analysis of the hemostatic, analgesic and healing effects of cyanoacrylate on free gingival graft surgical wounds in donor and recipient areas: a systematic review. J Mater Sci Mater Med. 2021 Aug 18;32(9):98. doi: 10.1007/s10856-021-06573-z. PMID 34406492